CLINICAL TRIAL: NCT05534074
Title: University Hospital of Ioannina COVID-19 Registry. Retrospective Datasource Registry of COVID-19 (Coronavirus Disease 2019) Hospitalized Patients
Brief Title: University Hospital of Ioannina COVID-19 (Coronavirus Disease 2019) Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Ioannina (Other)
Responsible Party: Principal Investigator, Liontos Angelos, Assistant Consultant of Internal Medicine, University Hospital, Ioannina
Other Study IDs: 4/21-4-2021 (Issue 24); 2022-003051-33 (EudraCT Number); U1111-1282-3362 (Other: World Health Organization, Universal Trial Number (UTN)); ΑΔΑ: Ψ29Ψ46906Η-9Τ0 (Other: Ministry of digital Governance of Greece); ΑΔΑ: Ψ29Ψ46906Η-9Τ0 (Other: diavgeia.gov.gr)
Record Dates: First submitted 2022-09-07; First posted 2022-09-09 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: COVID-19 (Coronavirus Disease 2019); COVID-19 Pandemic; COVID-19 Pneumonia; COVID-19 Respiratory Infection; COVID-19 Acute Respiratory Distress Syndrome; COVID-19-Associated Thromboembolism; COVID-19-Associated Pneumonia; COVID 19 Associated Coagulopathy
Keywords: COVID-19; SARS-CoV-2; COVID-19 registry
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVID-19 (Coronavirus Disease 2019) Registry of University Hospital of Ioannina. Retrospective datasource registry with quantitative and qualitative patient data from the hospital medical records. Epidemiological, clinical and laboratory parameters are recorded on 7 different time points (day: 1, 3, 5, 7, 9, 11, 15) concerning 793 variables of interest in an electronic (computerised) database. Patients are also followed-up after 90 days from hospital discharge (number of visits of follow-up depends on patient's health status) at the Post-COVID and Long-term effects of coronavirus (long COVID) outpatient clinic of University Hospital of Ioannina. Data from this outpatient clinic are also recorded in an electronic database (189 variables of concern for each patient)

DETAILED DESCRIPTION:
This is a retrospective study of COVID-19 (Coronavirus Disease 2019) at the Infectious Diseases Unit of the University Hospital of Ioannina. Quantitative and qualitative patient data are collected from the hospital medical records. Epidemiological, clinical and laboratory parameters are recorded on 7 different time points (day: 1, 3, 5, 7, 9, 11, 15) concerning 793 variables of interest in an electronic (computerised) database. Patients are also followed-up after 90 days from hospital discharge (number of visits of follow-up depends on patient's health status) at the Post-COVID and Long-term effects of coronavirus (long COVID) outpatient clinic of University Hospital of Ioannina. Data from this outpatient clinic are also recorded in an electronic database (189 variables of concern for each patient) The investigators collect data from COVID-19 hospitalized patients in the Infectious Diseases Unit of the University Hospital of Ioannina, from March 1st 2020 and ongoing. Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infection was diagnosed by reverse real time transcription-polymerase chain reaction (RT-PCR) test performed on nasopharyngeal swab specimens. Data are obtained retrospectively using patients' medical records (hard copy and digital records). All medical records are imported in a digital database anonymously with a personal identifier code for each patient, as prespecified by study protocol.

All data are collected following the highest standards set by the respective European Guidelines for Good Clinical and Laboratory Practice in Research Studies/Protocols and in accordance with the Helsinki Declaration. All participants in the study receive a personal identifier code and are kept anonymous. The epidemiological, clinical and laboratory data are collected and stored without being linked to personal data of the patients, but only to the personal identifier code. Biological samples are not collected. The collected clinical and laboratory data are archived in electronic databases (793 variables of concern for each individual patient).

ELIGIBILITY:
Inclusion Criteria:

* PCR positive for SARS-CoV-2
* hospitalization for COVID-19 disease in the Infectious Diseases Unit of University Hospital of Ioannina, greece

Exclusion Criteria:

* none

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: COVID-19 hospitalized patients
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
association of indices of COVID-19 severity with outcomes | 5 years
  outcomes: respiratory failure, disease severity in CT, death, intubation, length of stay

CONTACTS AND LOCATIONS:
Locations (1):
- 1st Division of Internal Medicine and Infectious Diseases Unit, University Hospital of Ioannina, Ioannina, Epirus, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Approval of the COVID-19 Registry from Administrative Board, Scientific Council, Ethics Committee and Research Committee of University Hospital of Ioannina, Greece — https://diavgeia.gov.gr/decision/view/%CE%A829%CE%A846906%CE%97-9%CE%A40